CLINICAL TRIAL: NCT00649142
Title: Prospective Study of Predisposing Factors for Chronic Postherniotomy Pain
Brief Title: Predisposing Factors for Chronic Postherniotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aesculap AG (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Henrik Kehlet, Professor, Ph D, M.D., Rigshospitalet, Section For Surgical Pathophysiology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: (KF) 01 294867
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Postherniotomy Pain
Keywords: Groin hernia; Chronic postsurgical pain; open mesh repair; laparoscopic mesh glue fixation; Sensory changes after groin hernia repair
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Open sutured mesh repair
  Interventions: Procedure: Open sutured mesh repair
- B (Active Comparator): Laparoscopic mesh glue fixation
  Interventions: Procedure: Laparoscopic mesh glue fixation

INTERVENTIONS:
Procedure: Open sutured mesh repair — Open sutured mesh repair
  Arms: A
Procedure: Laparoscopic mesh glue fixation — Laparoscopic mesh glue fixation
  Arms: B

SUMMARY:
Chronic pain affects pain in 5-8% of patients more than a year after groin hernia repair. However no prospective study has investigated potential predisposing factors for development of pain, including genetic, psychosocial and detailed neurophysiological assessment of surgical method.

The current study will assess the above factors in a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* Male
* Primary unilateral groin hernia
* Ability to use pain scales

Exclusion Criteria:

* Neurological disease
* Diabetes with late stage complications

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Frequency of chronic pain | 6 months postoperatively

SECONDARY OUTCOMES:
Changes in sensory function | 6 months
Influence of genotype, preoperative pain, intraoperative findings, psycho-social factors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, Professor, Ph D, M.D, Study Chair — Rigshospitalet, Copenhagen, section for surgical pathophysiology; Reinhard Bittner, Prof. Ph D, M.D., Principal Investigator — Marienhospital Stuttgart, Viszeralchirurgie
Locations (2):
- Ambulatory Surgical Clinic, Hørshom Sygehus, Hørsholm, Denmark
- Marienhospital, Viszeralchirurgie, Stuttgart, Germany

REFERENCES:
- [Background] Aasvang E, Kehlet H. Surgical management of chronic pain after inguinal hernia repair. Br J Surg. 2005 Jul;92(7):795-801. doi: 10.1002/bjs.5103. PMID 15962258